CLINICAL TRIAL: NCT04597151
Title: Diet Education Among Colorectal Cancer Survivors in the Safety Net Setting: A Pilot Feasibility Study
Brief Title: Diet Education Program for Stage I-IV Colorectal Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 204511; NCI-2020-06808 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-10-14; First posted 2020-10-22 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2022-01

CONDITIONS: Stage I Colorectal Cancer AJCC v8; Stage II Colorectal Cancer AJCC v8; Stage IIA Colorectal Cancer AJCC v8; Stage IIB Colorectal Cancer AJCC v8; Stage IIC Colorectal Cancer AJCC v8; Stage III Colorectal Cancer AJCC v8; Stage IIIA Colorectal Cancer AJCC v8; Stage IIIB Colorectal Cancer AJCC v8; Stage IIIC Colorectal Cancer AJCC v8; Stage IV Colorectal Cancer AJCC v8; Stage IVA Colorectal Cancer AJCC v8; Stage IVB Colorectal Cancer AJCC v8; Stage IVC Colorectal Cancer AJCC v8
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive care (diet education) (Experimental): Patients attend group diet education sessions over 1.5-2 hours every 2 weeks (weeks 1, 3, and 5).
  Interventions: Dietary Supplement: Dietary Intervention

INTERVENTIONS:
Dietary Supplement: Dietary Intervention — Attend diet education sessions
  Other Names: Dietary Modification; intervention, dietary; Nutrition Intervention; Nutrition Interventions; Nutritional Interventions

SUMMARY:
This pilot trial evaluates the feasibility of a group diet education program for stage I-IV colorectal cancer survivors. Providing a nutrition education program for colon and rectal cancer survivors may help them have better access to the tools necessary to make healthy food decisions that can impact their cancer outcomes.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To describe the feasibility and acceptability of a group diet education intervention for colorectal cancer (CRC) survivors at Zuckerberg San Francisco General Hospital (ZSFGH).

SECONDARY OBJECTIVE:

I. To describe perceived barriers to healthy diet among CRC survivors at ZSFGH.

EXPLORATORY OBJECTIVES:

I. To evaluate for differences in feasibility and acceptability of a group diet education program, based on sociodemographic factors such as education, food insecurity, employment, and race.

II. To explore changes in health-related behaviors pre and post intervention using a validated lifestyle score.

OUTLINE:

Patients attend group diet education sessions over 1.5-2 hours every 2 weeks (weeks 1, 3, and 5).

After completion of study, patients are followed up at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Able to speak and read English or Spanish
* Diagnosed with stage 1- 4 colorectal cancer within 5 years prior to study enrollment and treated with curative intent
* Receiving survivorship follow up care at Zuckerberg San Francisco General Hospital (ZSFGH)
* Able to provide written consent

Exclusion Criteria:

* Currently receiving chemotherapy, biologic therapy, radiation, or immunotherapy for colorectal cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Percentage of participants missing questionnaires | Up to 17 weeks
  Feasibility of measurement tools will be assessed by reporting the percentage of participants whom did not complete the questionnaires
Follow-up response rates | Up to 17 weeks
  Feasibility of measurement tools will be assessed by follow up response rates (week 6 and week 17)
Frequency of reasons for not participating in questionnaires | Up to 17 weeks
  Feasibility of measurement tools will be assessed by recording and reporting reasons for not taking part in questionnaires.
Number of participants who consent or expressed interest | Up to 17 weeks
  Subject recruitment will be assessed by number of participants who consent/number of participants who initially expressed interest, and reasons for non-participation will be documented.
Percentage of consented patients who remain on the study | Up to 17 weeks
  Subject retention will be assessed by percentage of consented patients who remain on the study at week 6 and at week 17, and reasons for dropout will be documented.
Number of sessions attended | Up to 17 weeks
  Adherence to diet education intervention will be assessed by number of sessions attended and reasons for absence will be documented.
Categorical responses to program evaluation survey | Up to 17 weeks
  Experience (e.g. satisfaction) will be assessed by tabulated responses to program evaluation survey. Qualitative analysis of cleaned and coded transcripts from interviews using a "constant comparison" process through which data are built into conceptual categories and themes will be performed.

SECONDARY OUTCOMES:
Frequency of responses to the baseline socio-demographics survey | Up to 17 weeks
  Barriers to healthy diet will be described using tabulated responses to the baseline socio-demographics survey and qualitative analysis of coded transcripts from baseline and exit interviews.

OTHER OUTCOMES:
Change in Lifestyle Score on the National Institute of Health (NIH)/ National Cancer Institute (NCI) Automated Self- Administered 24-hour Dietary Assessment Tool (ASA24) | Up to 17 weeks
  The ASA24® Dietary Assessment Tool is a free, web-based tool that enables multiple, automatically coded, self-administered 24-hour diet recalls and/or single or multi-day food records, also known as food diaries. The ASA24 system consists of a respondent website used to collect dietary intake data and a researcher website used to manage study logistics and obtain nutrient and food group data files to obtain analysis files for 65 nutrients and 37 food groups. This data is used to generate a standardized lifestyle score pre- and post-intervention with possible range: 0-7, based on participant's body mass index and intake of fruits and vegetables, fiber, ultra-processed foods, red meat, processed meat, sugar-sweetened drinks, and alcohol. This standardized score quantifies the degree to which participants' lifestyles are consistent with the 2018 World Cancer Research Fund (WCRF) / American Institute of Cancer Research (AICR) Recommendations.

CONTACTS AND LOCATIONS:
Overall Officials: Sorbarikor Piawah, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No